CLINICAL TRIAL: NCT06363045
Title: Comparative Study of the NIDEK TONOREF III with the Haag-Streit, Perkins Hand-held Applanation Tonometer for Tonometry Function and NIDEK TONOREF III with the NIDEK CEM-530 for Pachymetry Function
Brief Title: Comparative Study of the NIDEK TONOREF III with Predicate Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIDEK-TONOREF-UK-0001
Record Dates: First submitted 2024-03-24; First posted 2024-04-12 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults 18 years old or older (Experimental): NIDEK TONOREFIII
  Interventions: Device: NIDEK TONOREF III; Device: Haag-Streit, PERKINS HAND-HELD APPLANATION TONOMETER; Device: NIDEK CEM-530

INTERVENTIONS:
Device: NIDEK TONOREF III — The auto ref/kerato/tono/pachymeter TONOREF III is a medical device which measures objective refractive errors, corneal curvature radius, intraocular pressure and corneal thickness of the patient's eye.
Device: Haag-Streit, PERKINS HAND-HELD APPLANATION TONOMETER — Haag-Streit Goldmann Manual Tonometer measures intraocular pressure to aid in the screening and diagnosis of glaucoma
Device: NIDEK CEM-530 — Nidek CEM-530 is a non-contact ophthalmic microscope, optical pachymeter, and camera used for examination of the corneal endothelium and for measurement of the thickness of the cornea.

SUMMARY:
The primary objective of this clinical study is to prove that tonometry values for NIDEK TONOREF III are comparable to the predicate device and to prove that the pachymeter function of NIDEK TONOREF III is equivalent to the predicate device. The secondary objective is to demonstrate that the test device is as safe as the predicate devices.

ELIGIBILITY:
Exclusion criteria

1. Subjects with only one functional eye;
2. Those with one eye having poor or eccentric fixation;
3. Those with corneal scarring or who have had corneal surgery including corneal laser surgery;
4. Microphthalmos;
5. Buphthalmos;
6. Contact lens wearers;
7. Dry eyes;
8. Lid squeezers - blepharospasm;
9. Nystagmus;
10. Keratoconus;
11. Any other corneal or conjunctival pathology or infection.
12. central corneal thickness greater than 0,600 mm or less than 0,500 mm (2 standard deviations about the human mean)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Equivalent to legally-marketed devices | One or two study visits per subject. One visit is less than two hours.
  Agreement of intraocular pressure (mmHg) measurement for TONOREFIII and PAT
Equivalent to the pachymeter function | One or two study visits per subject. One visit is less than two hours.
  Agreement of central corneal thickness (µm) measurement for TONOREF III and CEM-530

SECONDARY OUTCOMES:
The numbers of adverse events | One or two study visits per subject. One visit is less than two hours.
  To demonstrate that the test device is as safe as the predicate devices.

CONTACTS AND LOCATIONS:
Overall Officials: Tadakazu Ichimura, Study Director — Nidek Co. LTD.
Locations (1):
- Aston University, Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No